CLINICAL TRIAL: NCT06541756
Title: Fibrine Clot-augmented Repair of Longitudinal Meniscus Tears - A Prospectively Randomized Controlled Trial
Brief Title: Fibrine Clot-augmented Repair of Longitudinal Meniscus Tears
Acronym: FCAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Collaborators: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Enejd Veizi, MD, Assistant Professor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2-24-7900
Record Dates: First submitted 2024-08-01; First posted 2024-08-07 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Meniscus Tear; Meniscus Lesion; Fibrin Blood Clot; Knee Injuries
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Controlled Study
Masking Description: not possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibrin Clot-augmented group (Experimental): Patients in the experimental repair group will undergo routine meniscus repair surgery in addition to a fibrin clot placed within the ruptured sides using arthroscopic all-inside or inside-out sutures. The fibrin clot will be prepared from 50cc of bone marrow aspirate obtained from the iliac crest and mixed for 15 minutes. The clot will be shaped into a cylindrical form and compressed between the torn edges of the meniscus using a trocar system, then secured with sutures.
  Interventions: Procedure: Fibrine Clot-augmented Meniscal Repair
- Conventionally repaired group (Active Comparator): Patients in the control repair group will undergo routine meniscus repair surgery using arthroscopic all-inside or inside-out sutures. The ruptured sides will be approximated as usual and the procedure will be considered completed.
  Interventions: Procedure: Conventional Meniscal Repair

INTERVENTIONS:
Procedure: Fibrine Clot-augmented Meniscal Repair — The fibrin clot will be prepared from 50cc of bone marrow aspirate obtained from the iliac crest and mixed for 15 minutes. The fibrin clot will be shaped into a cylindrical form and compressed between the torn edges of the meniscus using a trocar system, then secured with sutures.
  Arms: Fibrin Clot-augmented group
Procedure: Conventional Meniscal Repair — Patients in the standard repair group will undergo routine meniscus repair surgery using arthroscopic all-inside or inside-out sutures.
  Arms: Conventionally repaired group

SUMMARY:
Longitudinal meniscal tears are a type of meniscal injury characterized by a displaced fragment of the meniscus that flips over into the joint, often resembling a buckle or handle. These tears typically occur in the medial meniscus and are often associated with traumatic knee injuries, particularly in athletes.

The displaced meniscal fragment can cause mechanical symptoms such as locking, clicking, or catching of the knee, as well as pain and swelling. If not properly treated, buckle-handle meniscal tears can lead to further complications, including chronic knee instability, increased risk of osteoarthritis, and persistent joint pain.Repairing a longitudinal meniscal tear offers several advantages over partial meniscectomy, particularly in preserving knee function and preventing long-term complications.

Meniscal repair aims to restore the integrity of the meniscus, which plays a crucial role in load distribution, shock absorption, and joint stability.

Utilizing a fibrin clot during the repair of a buckle-handle meniscal tear can enhance the healing process and improve surgical outcomes. Fibrin clots act as a biological scaffold, promoting tissue regeneration by providing a matrix that facilitates cellular migration and proliferation.

The purpose of this study was to compare longitudinal meniscal tear repair reinforced with fibrin clot with routine end-to-end repair in a prospective randomized controlled trial.

DETAILED DESCRIPTION:
This study is designed as a prospective randomized controlled clinical trial. It aims to include patients presenting to the Orthopedics and Traumatology clinics at Ankara Bilkent and Etlik City Hospitals with longitudinal meniscus tears between August 2024 and December 2028. Participants will be randomly assigned to one of two groups: one receiving meniscus repair with fibrin clot reinforcement and the other receiving standard repair.

Patients in the standard repair group will undergo routine meniscus repair surgery using arthroscopic all-inside or inside-out sutures, with spinal anesthesia. For the fibrin clot group, a fibrin clot will be prepared from 50cc of bone marrow aspirate obtained from the iliac crest and mixed for 15 minutes. The fibrin clot will be shaped into a cylindrical form and compressed between the torn edges of the meniscus using a trocar system, then secured with sutures. After completing the repairs, the surgical wounds and portals will be closed, and an elastic bandage will be applied. The post-operative rehabilitation protocols will be the same for all patients.

Patients will be clinically followed for at least one year, with healing rates compared using control magnetic resonance imaging at the end of the first year.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with a painful meniscus (lateral or medial) longitudinal tear
* Being between the ages of 18 and 50
* Not having undergone surgery on the same knee before
* Having an MRI taken at the end of the 1st year post-surgery

Exclusion Criteria:

* Having additional collateral ligamentous damage along with the meniscus tear (such as MCL or LCL)
* Incomplete clinical scores at the end of the study
* A history of previous surgery on the same knee
* Having an active infection
* Not having a control MRI at the end of the 1st year

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with a healed meniscus on MRI | Postoperative 1st year
  Meniscal healing at 1 year follow up as detected on the control MRI (yes / no / partial)

SECONDARY OUTCOMES:
Tegner Activity Scale | Postoperative 1.st year
  minimum value:0, maximum value 10, higher values mean better outcome
The Knee injury and Osteoarthritis Outcome Score (KOOS) | Postoperative 1.st year
  minimum value:0, maximum value 100, higher values mean better outcome
Tegner-Lysholm Score | Postoperative 1.st year
  minimum value:0, maximum value 100, higher values mean better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Enejd Veizi, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Bilkent City Hospital, Ankara
  - Ankara Etlik City Hospital, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keller RE, O'Donnell EA, Medina GIS, Linderman SE, Cheng TTW, Sabbag OD, Oh LS. Biological augmentation of meniscal repair: a systematic review. Knee Surg Sports Traumatol Arthrosc. 2022 Jun;30(6):1915-1926. doi: 10.1007/s00167-021-06849-5. Epub 2022 Mar 8. PMID 35258647
- [Background] Chrysanthou C, Laliotis N, Paraskevas GK, Anastasopoulos N, Packer G. Enhancing Meniscal Repair: Investigating the Impact of an Exogenous Fibrin Clot. Cureus. 2024 Jan 27;16(1):e53083. doi: 10.7759/cureus.53083. eCollection 2024 Jan. PMID 38288322
- [Background] Rodriguez AN, Reist H, Liechti DJ, Geeslin AG, LaPrade RF. Shuttling Technique for Directed Fibrin Clot Placement During Augmented Inside-Out Repair of Horizontal Meniscus Tears. Arthrosc Tech. 2022 Nov 17;11(12):e2205-e2211. doi: 10.1016/j.eats.2022.08.027. eCollection 2022 Dec. PMID 36632380
- [Background] Kinoshita T, Hashimoto Y, Orita K, Iida K, Takahashi S, Nakamura H. Bone Marrow-Derived Fibrin Clots Stimulate Healing of a Knee Meniscal Defect in a Rabbit Model. Arthroscopy. 2023 Jul;39(7):1662-1670. doi: 10.1016/j.arthro.2022.12.013. Epub 2022 Dec 24. PMID 36574822
- [Background] Kale S, Deore S, Gunjotikar A, Singh S, Ghodke R, Agrawal P. Arthroscopic meniscus repair and augmentation with autologous fibrin clot in Indian population: A 2-year prospective study. J Clin Orthop Trauma. 2022 Aug 6;32:101969. doi: 10.1016/j.jcot.2022.101969. eCollection 2022 Sep. PMID 36035781